CLINICAL TRIAL: NCT05654272
Title: Development of Cardiovascular Innovation Research Technologies
Brief Title: Development of CIRC Technologies
Acronym: CIRC
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Christopher Nguyen, Director of Cardiovascular Innovation Research Center, The Cleveland Clinic
Other Study IDs: 22-737
Record Dates: First submitted 2022-11-27; First posted 2022-12-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases; Heart Failure; Ischemic Heart Disease; Non-ischemic Cardiomyopathy; Valvular Heart Disease; Metabolic Cardiomyopathy; Congenital Heart Disease; Aortic Diseases; Atrial Fibrillation; Ventricular Fibrillation
Keywords: MRI
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Myocardial Ischemia; Heart Valve Diseases; Heart Defects, Congenital; Aortic Diseases; Atrial Fibrillation; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: Normal volunteers >=18 years older
  Interventions: Diagnostic Test: MRI
- Cardiovascular Disease Patient: >=18years older with known prior cardiovascular disease
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Cardiac MRI

SUMMARY:
Cardiovascular disease is the leading cause of death worldwide. Advanced cardiovascular imaging using Magnetic Resonance Imaging (MRI) has proven to be effective in providing gold standard myocardial tissue characterization. Moreover, the intrinsic advantage of MRI's lack of exposure to ionizing radiation is particularly beneficial. At the same time, blood work can be very useful in early detection of certain cardiomyopathy, such as amyloid. However, there is a lack of agreement of on which markers are the most sensitive. This multi-study will allow us the unique opportunity to form a more comprehensive understanding for various cardiovascular diseases.

Our team has developed novel cardiac MRI techniques that leverages endogenous tissue properties to reveal a milieu of deep tissue phenotypes including myocardial inflammation, fibrosis, metabolism, and microstructural defects. Among these phenotypes, myocardial microstructure has proven to be most sensitive to early myocardial tissue damage and is predictive of myocardial regeneration. In this study, the investigators aim to further study the importance of cardiac microstructure revealed by MRI in patient and healthy population and compare this novel technology with conventional clinical biomarkers.

DETAILED DESCRIPTION:
The primary clinical objective of the clinical study is to determine and compare cardiac microstructural phenotypes by cardiac MRI in patients and healthy controls and their relationship to cardiac structure/function with our MRI technologies.

Aim 1: What are the myocardial microstructure phenotypes in both patients with cardiovascular disease and healthy cohorts? Are they linked to other prevalent macro structure and functional abnormalities?

The hypothesis is that the investigators can develop the next generation cardiac MRI exam that is faster, more robust, and more efficient for clinic use.

The enrolled subjects will do ONE of the following:

• Receive an extended clinical cardiac MRI exam. An MRI is an imaging technique used in radiology to make an accurate picture of the body. In this study the investigators will be focusing on the heart. The participant's routine clinical cardiac MRI exam will be extended by up to 25 min to perform a truncated research cardiac MRI protocol. The extended clinical cardiac MRI will take approximately one hour in total. The investigators may review the medical records to follow-up their medical status up to 5 years after start of the study.

OR:

• Receive a research cardiac non-contrast MRI exam. An MRI is an imaging technique used in radiology to make an accurate picture of the body. In this study the investigators will be focusing on the heart. The research cardiac MRI will take approximately one to two hours in total. The investigators may review the medical records to follow-up their medical status up to 5 years after start of the study

Optionally, if the subjects agree, the blood samples will be collected:

• Give blood sample for research purpose only. The blood draw is used to correlate the clinical blood biomarkers to the cardiac MRI data to help us better understand and validate the clinical utility of the novel cardiac MRI techniques. The blood draws should approximately take 20 minutes. The blood draw will take place in the doctor's office or at Mellen center private preparation by a registered nurse or approved technician. The blood will be stored with a unique code at Cleveland Clinic BioRepository for up to 10 years, and disposed following Cleveland Clinic guidelines. It may be used for future research in the Cleveland Clinic. Only members of the research team will have access to the participant's samples.

For healthy control:

• Only one cardiac MRI is needed, and it will be non-contrast MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Provision of written informed consent
* If not healthy volunteer, must be diagnosed with cardiovascular disease

Exclusion Criteria:

* Vulnerable populations will be excluded from this study including Prisoners
* Other contraindications to CMR imaging to be determined by standard MRI protocols
* Decisionally impaired (e.g., dementia or cognitive disability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of approximately 1000 eligible subjects either with cardiovascular disease or are healthy subjects. The investigators plan to enroll 800 patients and 200 healthy controls.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2032-09-09 (Estimated); Study Completion 2042-09-09 (Estimated)

PRIMARY OUTCOMES:
Myocardial Microstructure (Helix Angle) via Next Generation Cardiac MRI | 20 years
  The primary clinical objective of the clinical study is to determine and compare cardiac microstructural phenotypes by cardiac MRI in patients and healthy controls
Myocardial Function (Ejection Fraction) via Conventional Cardiac MRI | 20 years
  Measure cardiac function with conventional cardiac MRI to compare with other primary outcome of microstructure

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Innovation Research Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No